CLINICAL TRIAL: NCT05422300
Title: A 'Non-Invasive' Breath Test to Determine Anabolic Sensitivity in Females
Acronym: FBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FBT
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Dietary Protein; Female Protein Metabolism; Anabolic Sensitivity; Resistance Exercise; Young Adult Females
Keywords: Dietary Proteins/Administration & Dosage; Skeletal Muscle Metabolism; Human Adult Females; Diet; Exercise; Resistance Exercise; Amino Acids; Muscle Protein Synthesis; Skeletal Muscle Anabolism; Stable Isotopes
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study uses a 2-way counterbalanced crossover design. A total 10 young women (Ages: 18-35 years old) will be recruited and randomized into either the mid- follicular (7-10 days after the onset of menses) or mid-luteal phase (5-7 days after ovulation) (n=5, respectively). Participants will take part in two metabolic trials: Fed trial at rest (FED) and fed trial with resistance exercise (EX-FED). Following a minimum 3-day washout period, participants will complete the other trial, where both trials will be completed within the same phase of the menstrual cycle, depending on which group they were randomized into. Participants will be asked to self-report their menstrual cycle status, albeit ovulation test kits will be used to verify the cycle phase prior to each metabolic trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mid-Follicular Phase (Experimental): 7-10 days after the onset of menses, determined by self-reports and confirmed with ovulation test kits.
  Interventions: Behavioral: Fed; Behavioral: Ex-Fed
- Mid-Luteal Phase (Experimental): 5-7 days after ovulation, determined by self-reports and confirmed with ovulation test kits.
  Interventions: Behavioral: Fed; Behavioral: Ex-Fed

INTERVENTIONS:
Behavioral: Fed — Subjects will be fed a mixed-macronutrient beverage at rest (0.75g/kg lean body mass of carbohydrates; 0.25g/kg lean body mass of protein). Amino acid composition of the protein will be modelled off the composition of egg. Leucine content will be enriched to 5% with [13C]-leucine.
  Other Names: Feeding at Rest
Behavioral: Ex-Fed — Participants will be subjected to a full-body resistance exercise protocol, consisting of an upper and lower body circuit. The upper body circuit will be a chest press and dumbbell row superset, whereas the lower body circuit will be leg press and leg extension (4 sets of 10 repetitions @ 75% of their 1 repetition max, respectively). The inter-set rest period will be 90 seconds.
  Subjects will be fed a mixed-macronutrient beverage at rest (0.75g/kg lean body mass of carbohydrates; 0.25g/kg lean body mass of protein). Amino acid composition of the protein will be modelled off the composition of egg. Leucine content will be enriched to 5% with [13C]-leucine.
  Other Names: Exercise with Feeding

SUMMARY:
The maintenance of lean body mass, especially skeletal muscle, is vital for optimal health and performance across the lifespan. The protein component of lean body mass is in a constant state of turnover, involving the simultaneous breakdown of old and/or damaged proteins and the synthesis of new proteins. These processes collectively determine if someone gains or loses lean body mass. Eating a protein-rich meal or performing resistance exercise can stimulate protein synthesis to gain lean body mass. Stable isotope "tracers" are amino acid building blocks that are slightly heavier than those naturally found in the body. In research, these are often used to assess changes in protein turnover in response to feeding and/or exercise. However, traditional stable isotope tracer methods involve the intravenous delivery of a tracer with blood sampling and muscle biopsies, which may be cumbersome or unfeasible for some for participants.

The investigators have recently developed and validated a non-invasive 'breath test' in males that measures the efficiency of the body for using amino acids in food to build new body proteins. The principle of this method is that leucine, an essential amino acid that the body must acquire from normal diet, can be used to build new body proteins or as a source of energy (i.e., oxidized). Since leucine is preferentially used in skeletal muscle, skeletal muscle protein metabolism can be non-invasively inferred . Any leucine "tracer" that is oxidized can be detected and measured in the carbon dioxide exhaled. It has been observed that less dietary leucine is oxidized when active males perform a bout of resistance exercise, meaning more was used to build muscle proteins. When performed habitually, resistance exercise can help skeletal muscles grow, compared to a rested-state, resulting in greater leucine retention in the body to build new proteins. Therefore, the purpose of this study is to validate this non-invasive breath test in females to increase the validity of the method in a wider range of populations. Ultimately, the results will further validate this non-invasive tool that can potentially detect whether different populations are sensitive to dietary amino acids and in a position to gain or lose lean body mass.

DETAILED DESCRIPTION:
The objective of the present study is to validate the use of an oral L-[13C]-leucine stable isotope tracer, preferentially metabolized within skeletal muscle, to detect an exercise-induced increase in anabolic sensitivity (i.e., reduction in oxidation) in females. It is hypothesized that since resistance exercise enhances skeletal muscle protein synthesis, anabolic sensitivity measured through leucine retention would be greater with feeding after resistance exercise compared to feeding at rest.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* 18-35 years of age
* BMI ≥18.5 kg/m2 and ≤ 30 kg/m2
* Eumenorrheic (self-reported menstruation for prior 3 consecutive months)
* Recreationally active; currently performing structured exercise (e.g. running, weightlifting, team-sport activity) at least once per week for ≥ 6 months before enrolment

Exclusion Criteria:

* Use of oral contraceptives
* Inability to perform physical activity as determined by the PAR-Q+
* Inability to adhere to protocol guidelines (e.g. alcohol, caffeine, habitual diet)
* Regular tobacco use
* Illicit drug use (e.g. growth hormone, testosterone, etc...)
* Diagnosed medical condition under the care of a physician (e.g. type 2 diabetes)
* Inability to abstain from supplements (e.g. protein, creatine, HMB, BCAA, phosphatidic acid, etc...) at least three weeks before the trial
* Individuals on any medications known to affect protein metabolism (e.g. corticosteroids, non-steroidal anti-inflammatories, and/or prescription-strength acne medications)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Net-Leucine Retention (umol/kg) | 6 hours
  Whole-Body Net Leucine Retention determined from the difference between exogenous leucine oxidation and leucine ingestion the 6 hour measurement period.
Exogenous Leucine Oxidation (umol/kg) | 6 hours
  Exogenous Leucine Oxidation determined from breath 13CCO2 enrichment. Breath samples will be collected every 20-30min after test drink ingestion to determine breath 13CO2 enrichment. Total leucine oxidation will be determined from the area under the 13CO2 enrichment by time curve.

CONTACTS AND LOCATIONS:
Overall Officials: Nicki Pourhashemi, MSc Student, Study Director — Faculty of Kinesiology and Physical Education; Hugo JW Fung, PhD (c), Study Director — Faculty of Kinesiology and Physical Education; Jonathan Aguilera, PhD Student, Study Director — Faculty of Kinesiology and Physical Education
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No